CLINICAL TRIAL: NCT05492877
Title: A Phase IIa Randomised, Double Blind, Placebo Controlled, Parallel Arm, Multi-Centre Study to Evaluate the Efficacy and Safety of Mitiperstat (AZD4831), for 12-24 Weeks, in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: An Efficacy and Safety Study of Mitiperstat (AZD4831) (MPO Inhibitor) vs Placebo in the Treatment of Moderate to Severe COPD.
Acronym: CRESCENDO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6582C00001; 2022-002441-18 (EudraCT Number)
Record Dates: First submitted 2022-07-22; First posted 2022-08-09 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Mitiperstat; AZD4831; Myeloperoxidase; MPO; Myeloperoxidase inhibitor; COPD; Chronic Obstructive Pulmonary Disease; Lung function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — AZD4831

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to receive either Mitiperstat (AZD4831) or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Approximately 203 participants will be randomised to receive placebo.
  Interventions: Other: Placebo
- Mitiperstat (AZD4831) (Experimental): Approximately 203 participants will be randomised to receive mitiperstat (AZD4831).
  Interventions: Drug: Mitiperstat (AZD4831)

INTERVENTIONS:
Drug: Mitiperstat (AZD4831) — Oral dosage, once daily.
  Arms: Mitiperstat (AZD4831)
Other: Placebo — Oral dosage, once daily.
  Arms: Placebo

SUMMARY:
This is a research study to evaluate the efficacy and safety of the investigational drug Mitiperstat (AZD4831) in adult patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Study D6582C00001 is a phase IIa randomised, double blind, placebo controlled, parallel arm study to evaluate the efficacy and safety of Mitiperstat (AZD4831) in adult participants with moderate to severe chronic obstructive pulmonary disease.

Approximately 100 sites globally will participate in this study. Approximately 406 participants will be randomised to two treatment groups; Mitiperstat (AZD4831) vs placebo in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent.
* Participants must be deemed as high risk of exacerbations as defined by: >= 1 moderate or severe exacerbation in the previous 24 months; or frequent productive cough; or post-bronchodilator (BD) forced expiratory volume in the first second (FEV1) < 50% predicted.
* Participants must be 40-80 years of age inclusive, at the time of signing informed consent form (ICF).
* Participants who have a confirmed primary diagnosis of moderate to severe COPD.
* Participants who are current or ex-smokers with a tobacco history of ≥ 10 pack-years.
* Participants who have a documented stable regimen of triple therapy or dual therapy for

  ≥ 3 months prior to enrolment.
* Body mass index within the range 18 to 40 kg/m2 (inclusive).

Exclusion Criteria:

* As judged by the investigator, any evidence of any active medical or psychiatric condition or other reason (at SV1 [screening] and SV3 [pre-dose]) which in the investigator's opinion makes it undesirable for the participant to participate in the study.
* Current diagnosis of asthma or past diagnosis of asthma which persisted beyond the age of 25 years.
* Clinically important pulmonary disease other than COPD.
* Any other clinically relevant abnormal findings on physical examination, laboratory testing including haematology, coagulation, serum chemistry, or urinalysis; or chest CT scan at screening or randomisation, which in the opinion of the investigator or medical monitor may compromise the safety of the participant in the study or interfere with evaluation of the study intervention or reduce the participant's ability to participate in the study.
* History of a clinically significant infection (viral, bacterial, or fungal; defined as requiring systemic antibiotics, antiviral, or antifungal medication for > 7 days) within 4 weeks prior to SV3 (Day 1) (including unexplained diarrhoea) or clinical suspicion of infection at time of dosing.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (93):
- United States (19):
  - Research Site, Newport Beach, California
  - Research Site, Clearwater, Florida
  - Research Site, DeLand, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Chicago Ridge, Illinois
  - Research Site, Ann Arbor, Michigan
  - Research Site, Chesterfield, Missouri
  - Research Site, Saint Charles, Missouri
  - Research Site, New Windsor, New York
  - Research Site, Gastonia, North Carolina
  - Research Site, Kernersville, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Choctaw, Oklahoma
  - Research Site, Fort Mill, South Carolina
  - Research Site, Amarillo, Texas
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, Córdoba
  - Research Site, Ranelagh
  - Research Site, San Fernando
- Bulgaria (7):
  - Research Site, Dupnitsa
  - Research Site, Haskovo
  - Research Site, Pernik
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Vratsa
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Næstved
  - Research Site, Odense C
  - Research Site, Vejle
- Germany (8):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Immenhausen
  - Research Site, Koblenz
  - Research Site, Landsberg
  - Research Site, Leipzig
  - Research Site, Marburg
  - Research Site, Witten
- Italy (5):
  - Research Site, Foggia
  - Research Site, Roma
  - Research Site, Sassari
  - Research Site, Siena
  - Research Site, Verona
- Mexico (5):
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Monterrey
  - Research Site, Veracruz
  - Research Site, Zapopan
- Netherlands (2):
  - Research Site, Groningen
  - Research Site, Veldhoven
- Poland (8):
  - Research Site, Bielsko-Biala
  - Research Site, Chęciny
  - Research Site, Karczew
  - Research Site, Krakow
  - Research Site, Ksawerów
  - Research Site, Staszów
  - Research Site, Szczecin
  - Research Site, Warsaw
- South Africa (4):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Tygervalley
  - Research Site, Vereeniging
- Spain (5):
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Mérida
  - Research Site, Santander
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Mersin
- United Kingdom (11):
  - Research Site, Bradford
  - Research Site, Cambridge
  - Research Site, Cottingham
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Rotherham
  - Research Site, Wakefield
  - Research Site, York

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: D6582C00001 CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6582C00001&attachmentIdentifier=9d47cf65-5b68-48b9-ad78-4cbf1f20dc73&fileName=D6582C00001_CSR_Synopsis.pdf&versionIdentifier=
- See also: D6582C00001 CSP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6582C00001&attachmentIdentifier=89f77e0b-c8f3-4846-ba7c-c06eff7c61b7&fileName=D6582C00001_CSP_Redacted.pdf&versionIdentifier=
- See also: D6582C00001 SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6582C00001&attachmentIdentifier=d65d77d3-86ba-4ff5-8216-8a79e4b1f09f&fileName=D6582C00001_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 101 centers in 14 countries (Argentina, Bulgaria, Canada, Denmark, Germany, Italy, Mexico, Netherlands, Poland, South Africa, Spain, Turkey, UK and USA).
Pre-assignment Details: A total of 381 participants were randomized and received at least one dose of study drug.
Groups:
- Mitiperstat: Participants received an oral tablet of mitiperstat 5mg once daily.
- Placebo: Participants receive an oral tablet of placebo matched to mitiperstat once daily.
Period: Overall Study
Arm/Group | Mitiperstat | Placebo
Started | 189 | 192
Treated | 189 | 192
Completed | 165 | 170
Not Completed | 24 | 22
Not completed — Adverse Event | 11 | 7
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Reason not specified | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mitiperstat | Placebo | Total
Number analyzed (Participants) | 189 | 192 | 381
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (6.65) | 65.7 (7.03) | 66 (6.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 74 | 151
  Male | 112 | 118 | 230
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 27 | 53
  Not Hispanic or Latino | 163 | 165 | 328
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 182 | 183 | 365
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Effect of Mitiperstat (AZD4831) as Compared to Placebo on the Time to First COPD Composite Exacerbation (CompEx) Event in Patients With Moderate to Severe COPD.
Description: COPDCompEx is a composite endpoint of exacerbations and events defined from participant e-Diaries and peak expiratory flow (PEF). COPDCompEx defined exacerbations included episodes leading to one or more of the following: hospitalization, emergency room visit, treatment with systemic corticosteroids (injected and/or oral), or treatment with antibiotics. Diary COPDCompEx events are defined by threshold and slope criteria being met for >= 2 consecutive days using the following diary and home spirometry variables: overall symptom rating, night-time awakenings due to symptoms, reliever medication use, PEF. COPDCompEx also includes patient withdrawals for treatment failure.
Time Frame: From baseline to up to 24 weeks
Population: Full Analysis Set (FAS) included all randomised participants who received at least one dose of study intervention. 'While on treatment' estimand strategy was followed, which means that if an intercurrent event occurs all subsequent data for that subject was excluded from the evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Mitiperstat | Placebo
Number analyzed (Participants) | 189 | 192
Participants | 125 | 125
Statistical Analysis 1: Comparison: Mitiperstat vs Placebo; Test type: Superiority; p = 0.599, Regression, Cox; Hazard Ratio (HR) = 1.071, 90% CI 2-sided [0.869 to 1.320]; The p-value was based on a 2-sided log rank test stratified by region

2. Secondary Outcome: To Assess the PK of Mitiperstat (AZD4831) in Patients With Moderate to Severe COPD
Description: Measurement of Time to Reach Maximum Plasma Concentration (Tmax) at pre-randomisation (baseline visit) and week 12.
Time Frame: At week 12
Population: The PK set included all participants who had received mitiperstat and had evaluable PK data for mitiperstat, with no important protocol deviations that were thought to have impacted the analysis of the PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Mitiperstat
Number analyzed (Participants) | 36
hours | 1.292 [0.42 to 2.92]

3. Secondary Outcome: To Assess the Pharmacokinetics (PK) of Mitiperstat (AZD4831) in Patients With Moderate to Severe COPD.
Description: Measurement of Maximum Plasma Concentration (Cmax) at pre-randomisation (baseline visit) and week 12.
Time Frame: At week 12
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Mitiperstat
Number analyzed (Participants) | 36
nmol/L | 38.786 (39.5)

4. Secondary Outcome: To Evaluate the Effect of Mitiperstat (AZD4831) as Compared to Placebo on the Time to First Moderate or Severe Exacerbation.
Description: A COPD exacerbation was considered moderate if it required treatment with systemic corticosteroids and/or antibiotics for at least 3 days or resulted in emergency room visit< 24 hours requiring intensive treatment; and did not result in hospitalization or death.
  A COPD exacerbation was considered severe if it resulted in hospitalization (defined as an inpatient admission ≥ 24 hours in the hospital, an observation area, the emergency department, or other equivalent healthcare facility depending on the country and healthcare system) or death due to COPD.
Time Frame: From baseline to up to week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mitiperstat | Placebo
Number analyzed (Participants) | 189 | 192
Participants | 53 | 44
Statistical Analysis 1: Comparison: Mitiperstat vs Placebo; Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 1.234, 90% CI 2-sided [0.882 to 1.726]

5. Secondary Outcome: To Assess the Effects of Mitiperstat (AZD4831) as Compared to Placebo on Post-bronchodilator (BD) Forced Expiratory Volume in the First Second (FEV1) in Patients With Moderate to Severe COPD.
Description: The mean change from baseline in Post-BD FEV1 at Week 12 was estimated using a repeated measures mixed effects analysis of covariance. Only subjects with non-missing covariates are included in the analysis. FEV1 was measured by spirometry at clinic.
Time Frame: From baseline to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Mitiperstat | Placebo
Number analyzed (Participants) | 130 | 136
Litre | -0.049 (0.0178) | -0.031 (0.0175)

6. Secondary Outcome: To Assess the Effect of Mitiperstat (AZD4831) Compared to Placebo on Respiratory Symptoms in Patients With Moderate to Severe COPD.
Description: Change from baseline in EXAcerbations of Chronic Pulmonary Disease Tool (EXACT) which is a 14-item ePRO instrument developed to assess the frequency, severity and duration of COPD exacerbations. It has a theoretical range of 0 to 100, with higher values indicating a more severe condition. The EXACT will be performed at on-site visits using the e-Diary.
Time Frame: From baseline to week 12 and week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Mitiperstat | Placebo
Number analyzed (Participants) | 122 | 126
Units on a scale
  Week 12: number analyzed (Participants) | 118 | 123
  Week 12 | 0.1 (0.97) | -2.4 (0.95)
  Week 24: number analyzed (Participants) | 54 | 50
  Week 24 | -1.9 (1.32) | -3.7 (1.36)

7. Secondary Outcome: To Assess the Effect of Mitiperstat (AZD4831) Compared to Placebo on Respiratory Symptoms in Patients With Moderate to Severe COPD.
Description: Change from baseline to Week 12 and week 24 in mean Breathlessness, Cough and Sputum Scale (BCSS) score is reported. The BCSS was a 3-item daily diary that assesses the severity of the 3 symptoms: breathlessness, sputum, and cough, each on a 5-point Likert scale ranging from 0 (no symptoms) to 4 (severe symptoms). Item scores were summed to yield a total score ranging from 0 to 12; wherein higher total score indicated more severe symptoms. The BCSS was captured each evening via eDiary.
Time Frame: From baseline to week 12 and week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Mitiperstat | Placebo
Number analyzed (Participants) | 139 | 147
Units on a scale
  Week 12: number analyzed (Participants) | 138 | 146
  Week 12 | 0.16 (0.130) | 0.15 (0.127)
  Week 24: number analyzed (Participants) | 71 | 63
  Week 24 | 0.11 (0.166) | -0.17 (0.172)

8. Secondary Outcome: To Assess the Effect of Mitiperstat (AZD4831) Compared to Placebo in Disease Impact in Patients With Moderate to Severe COPD.
Description: Change from baseline to Week 12 and week 24 in cough Visual Analogue Scale (VAS) score is reported. Participants were asked to complete a cough severity VAS (100-point linear scale marked with a horizontal line by the participant, with 0 representing ''no cough'' and 100 representing "worst cough") that measured subjective assessment by the participant of the prior 24 hrs for severity of cough symptoms. It was completed each evening in the eDiary.
Time Frame: From baseline to week 12 and week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Mitiperstat | Placebo
Number analyzed (Participants) | 159 | 165
Units on a scale
  Week 12: number analyzed (Participants) | 157 | 165
  Week 12 | -1.25 (1.183) | -3.05 (1.160)
  Week 24: number analyzed (Participants) | 81 | 73
  Week 24 | -2.64 (1.540) | -3.48 (1.562)

9. Secondary Outcome: Change From Baseline to Week 12 in Total COPD Assessment Test (CAT)
Description: COPD Assessment Test (CAT) is designed to measure how COPD impacts on a patient's daily life and how this might change over time. It consists of 8 questions that ask the patient to rate items relating to symptoms and impact on quality of life (such as normal activity and sleep). Each question is performed on a 5-point Likert scale from 0 (no symptoms/no impact) to 5 (severe symptoms/impact). The CAT will be completed by participants at on-site visits using the e-Diary.
Time Frame: From baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Mitiperstat | Placebo
Number analyzed (Participants) | 134 | 134
Units on a scale | -1.2 (0.62) | -1.2 (0.64)

ADVERSE EVENTS:
Time Frame: From Day 1 to Week 24
Arm/Group | Mitiperstat | Placebo
All-Cause Mortality (participants affected / at risk) | 1/189 | 0/192
Serious Adverse Events (participants affected / at risk) | 23/189 | 13/192
Other Adverse Events (participants affected / at risk) | 53/189 | 45/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitiperstat (N=189) | Placebo (N=192)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Carotid artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitiperstat (N=189) | Placebo (N=192)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 45 (62) | 36 (55)
Nasopharyngitis (Infections and infestations) | 11 (11) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT05492877/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT05492877/SAP_001.pdf